CLINICAL TRIAL: NCT04249609
Title: The Effect of Macronutrient Composition of Meals Consumed Around a Single Exercise Session of Subjective Appetite, Appetite Hormones and Daily Energy Intake in Overweight Men
Brief Title: Composition of Meals Around Exercise Session
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Dr Dalia Malkova Senior Lecture in Human Nutrition, School of Medicine, Dentistry & Nursing, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200180122
Record Dates: First submitted 2019-11-01; First posted 2020-01-31 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Hormones
Keywords: Exercise; Appetite; Gastrointestinal hormones; Macronutrient; Fat oxidation; Thermic effect of food; Energy intake
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Carbohydrate Meals Around Exercise (Experimental): On day 1, high CHO dinner meal will provide 35% of participants total daily energy requirements. Meal will consist of pasta, meat ball and orange juice. On the day 2, participants will exercise for 60 minutes and then in 60 minutes will consume morning meal, providing 30% of their total daily energy requirements. Morning meal will consist of oats, skimmed-milk, banana and seedless raisins.
  Interventions: Other: HCHO meals and exercise
- Low Carbohydrate Meals Around Exercise (Experimental): On day 1, low CHO dinner meal will provide 35% of participants total daily energy requirements. Meal will based on burger, cheese, mushroom, nuts, and butter.On the day 2, participants will exercise fro 60 minutes and then in 60 will consume morning meal, providing 30% of their total daily energy requirements. Meal will consist of white bread, egg, cheese, olive oil, nuts, and olives.
  Interventions: Other: LCHO meals and exercise

INTERVENTIONS:
Other: HCHO meals and exercise — Exercise will be conducted after high carbohydrate dinner and prior to high carbohydrate breakfast
  Other Names: High carbohydrate meals and exercise
  Arms: High Carbohydrate Meals Around Exercise
Other: LCHO meals and exercise — Exercise will be conducted after high fat dinner and prior to high fat breakfast
  Other Names: Low Carbohydrate and exercise Intervention
  Arms: Low Carbohydrate Meals Around Exercise

SUMMARY:
This will be a randomised cross-over study where participants will be asked to undergo screening session followed by submaximal exercise test and then undergo 2 experimental trials, one high CHO trial and another high fat trial, each lasting over 2 days. On Day 1 participants will consume either high CHO or high fat evening meal and on Day 2 they will be exercising for 60 minutes in the fasted state and then consume either high CHO or high fat morning meal and then 5 hours after morning meal ad libitum buffet meal. After this, they will leave metabolic investigation room and will record all food and drinks consumed during the rest of the day. The washout period between the trials will be at least 7 days. Prior to each of the experimental trials, participants will be asked to avoid consumption of coffee and alcohol for the duration of 2 days. All data collection will all take place in the metabolic research unit at New Lister Building (NLB), Glasgow Royal infirmary (GRI).

DETAILED DESCRIPTION:
The researcher will enrol eligible participants by means of an advertisement leaflet and word of mouth in the campus of the University of Glasgow and other major public areas. Those who show interest about the study will be contacted by the researcher who will explain the study in detail and will give them a copy of the participant information leaflet. If the participant is happy to participate, he will sign an informed consent form and privacy notes. Only participants with stable body weight for at least 3 months will be recruited and we will exclude those who are on positive or negative energy balance (recent weight gain or loss, ±2 kg the past month).

As part of the screening process, each participant will be asked to fill in Physical Activity Readiness Questionnaire (PARQ) and Health Screening Questionnaire. Only those who answered "no" to all questions in PARQ and were in generally good health will carry on with other aspects of the study. These questionnaires will be completed during screening session, which will take place at NLB, GRI. Height and body weigh will be measured at the screening session. Only those with BMI between 25.0-30 kg/m2 will be invited to participate. Smokers will not be recruited. It will be explained that their participation is voluntary, that they may withdraw at any point if they wish, and that the data collected will be anonymised. We will thank those subjects who have expressed an interest about the study but do not qualify and we will explain to them why they need to be excluded. Those who are eligible to participate will be enrolled in the trial which will last for 4 weeks and we will measure their height and weight.

Main Experimental Trials:

The experimental trials will last over 2 days. On day 1 Participants will consume provided dinner and on Day2 attend the metabolic research unit at New Lister Building of the Royal Infirmary in the fasted state at approximately 09:00 am. An intravenous cannula will be placed by a trained phlebotomist upon arrival. This will be used to draw blood samples throughout trial. After the collection of the first blood sample, the participant will walk on the treadmill at speed and grade corresponding to 55% of their maximal oxygen consumption. During exercise, participants will be wearing a heart rate monitor and a face mask connected to indirect calorimetry equipment to allow measurements of fat and CHO oxidation Ratings of perceived exertion will be recorded at every 10 minutes. Following exercise, participants will rest for 60 minutes and then either high CHO or high fat morning meal will be provided. Further blood samples will be collected for the duration of 5-hours; in total no more than 70 ml of blood will be taken during each of the trials. Following the last blood sample collection, participants will eat from ad libitum buffet and then leave laboratory and during the rest of the day will be recording all food and drink consumed.

Meal On day 1 dinner meal will provided with either high carbohydrate or high fat meal which contains 35% of participants total daily energy intakes. In high CHO trial, meal will consist of pasta, meat ball and orange juice. In high fat trial, meals will be based on burger, cheese, mushroom, nuts, and butter. On the day 2 and after 60 minutes exercise, participants will consume morning meal, providing 30% of their total daily energy intake. In high fat trial, morning meals will be based on white bread, peanut butter, nuts, and olives. In high CHO trial, meal will consist of oats, skimmed milk, banana and seedless raisins.

Exercise Tests Participants will conduct a submaximal exercise test to estimate their maximal oxygen consumption (V̇O2 max), a marker of cardiorespiratory fitness. During the main experimental trials, participants will undergo a 60-minute walking exercise at a predetermined work rate corresponding to 55% of their predicted V̇O2 max. Both exercise sessions will be conducted on a treadmill and will be at intensity below 85% of maximal HR. Heart rate and ratings of perceived exertion will be recorded throughout the test via a heart rate monitor.

Preparation for experimental trials Participants will be asked to record dietary intake for 2 days prior to the first experimental trial and will be asked to replicate this in the 2 days prior to the second experimental trial. Prior to both experimental trials participants will be asked to avoid consumption of coffee and alcohol for the duration of 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy sedentary males aged between 25-35 years with body mass index (BMI) 25- 30 kg/m2
* participants with stable body weight for at least 3 months.

Exclusion Criteria:

* Smokers, suffering from food allergy, on any dietary supplements or dietary regimes at the time of the study
* Participants with systolic/diastolic <90/60 mmHg and >140/90 mmHg or with history of chronic illness.

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Appetite Hormones: Glucagon like peptide (GLP-1) | 420 minutes through study completion, an average of 10 days
  Plasma concentration during HCHO and LCHO trials
Appetite Hormone: Peptide YY (PYY) | 420 minutes through study completion, an average of 10 days
  Plasma concentration during HCHO and LCHO trials
Growth Differentiation Factor-15 (GDF 15) | 420 minutes through study completion, an average of 10 days
  Plasma concentration during HCHO and LCHO trials

SECONDARY OUTCOMES:
Insulin | 420 minutes through study completion, an average of 10 days
  Plasma concentration during HCHO and LCHO trials
Glucose | 420 minutes through study completion, an average of 10 days
  Plasma concentration during HCHO and LCHO trials
Triglycerides | 420 minutes through study completion, an average of 10 days
  Plasma concentration during HCHO and LCHO trials
Subjective appetite scores | 420 minutes through study completion, an average of 10 days
  Appetite scores during HCHO and LCHO trials will be assessed using a 100-mm Visual Analog Scale, with 0 mm meaning one and 100 mm another extreme of hunger, desire to eat, fullness, prospective food consumption, and satiety.
Diet induced thermogenesis | 420 minutes through study completion, an average of 10 days
  Metabolic rate measured during HCHO and LCHO trials by means of indirect calorimetry
Dietary intake | 24 hr through study completion, an average of 10 days
  Energy and macronutrient intake during HCHO and LCHO trial will analyses using WinDiets software based on food composition tables.
Energy substrate oxidation | 420 minutes through study completion, an average of 10 days
  Rate of carbohydrate and fat oxidation during HCHO and LCHO trials by means of indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Malkova, PhD, Study Chair — University of Glasgow
Locations (1):
- Human Nutrition, College of Medicine, Veterinary and Life Science, Glasgow, United Kingdom